CLINICAL TRIAL: NCT02371655
Title: Different Bowel Preparations in CT Colonography: is Diet Necessary? A Randomized Controlled Trial
Acronym: DIETSAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Davide Bellini, Medical Doctor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: URomLSDBAL1
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Cathartic Colon; Colonic Neoplasms
Keywords: Bowel cleansing; CTcolonography; Bowel preparation; Faecal and fluid tagging
MeSH Terms: conditions — Colonic Neoplasms | interventions — Diet

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet included (Active Comparator): Diet is included in bowel preparation
  Interventions: Procedure: Diet; Drug: Faecal Tagging; Drug: Bowel cleansing; Procedure: CT colonography
- Diet not included (Experimental): Diet is not included in bowel preparation
  Interventions: Drug: Faecal Tagging; Drug: Bowel cleansing; Procedure: CT colonography

INTERVENTIONS:
Procedure: Diet — A low-fibre diet for three days before the examination
  Other Names: diet included
  Arms: Diet included
Drug: Faecal Tagging — Oral ingestion of iodinated contrast media (Gastrografin 60 ml) 3h before the examination
  Other Names: iodinated contrast media (oral)
Drug: Bowel cleansing — Oral ingestion of water solution (macrogol 100 mg, Sanipeg) the day before the examination
  Other Names: chatartic bowel preparation
Procedure: CT colonography — CT Examination of the colon aimed to detect polyps and cancer
  Other Names: Virtual colonoscopy

SUMMARY:
The aim of this study is to compare a new regimen of reduced bowel preparation that does not include low fiber diet with another reduced bowel preparation including low-fiber diet.

DETAILED DESCRIPTION:
Bowel preparation should be safe and well tolerated by patients, particularly in a screening setting. For this reason, limited bowel preparations have been extensively investigated. Usually, they combine the use of low-fibre diet and faecal/fluid tagging. The ingestion of a positive contrast agent (either barium, iodine or a combination of the two),needed to differentiate stool or fluid residues from true colonic lesions, is now considered mandatory. A low-fibre diet has the aim of improving residue homogeneity and facilitates tagging; however, there aren't significative evidences at support. The aim of this study is to compare a new regimen of reduced bowel preparation that does not include low fiber diet with another reduced bowel preparation including low-fiber diet. Primary outcome is the overall quality of bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients (Screening Patients)
* Symptomatic patients unwilling to undergo optical colonoscopy (Symptomatic Patients)
* Patients with a previous incomplete optical colonoscopy.

Exclusion Criteria:

* Allergy to Macrogol
* Cognitive behavioral deficits

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
overall quality of bowel preparation using a 0-3 scale for each parameter (Homogeneity of solid-fluid fecal tagging, volume of residual fluid, colon distension). | 1 day
  the evaluation of overall quality of bowel preparation on CT colonography images including: homogeneity of tagging, presence of unmarked solid stool residues, the evaluation of volume of residual fluids and colon distention.

SECONDARY OUTCOMES:
compliance of patients | 1 day
  A 0-10 visual analogical scale (VAS) was used with 0 corresponding to no discomfort and 10 to severe discomfort with severe impact on patient's daily activities. Intermediate values corresponded to intermediate values of tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Laghi Andrea, Professor, Study Director — University of Rome "Sapienza" Faculty of Medicine and Dentistry Department of Radiological Sciences, Oncology and Pathology I.C.O.T. - Via F. Faggiana 34, 04100 Latina, Italy
Locations (1):
- ICOT Hospital, Sapienza, Latina, Italy

REFERENCES:
- [Background] Liedenbaum MH, Denters MJ, de Vries AH, van Ravesteijn VF, Bipat S, Vos FM, Dekker E, Stoker J. Low-fiber diet in limited bowel preparation for CT colonography: Influence on image quality and patient acceptance. AJR Am J Roentgenol. 2010 Jul;195(1):W31-7. doi: 10.2214/AJR.09.3572. PMID 20566777
- [Background] Iafrate F, Iannitti M, Ciolina M, Baldassari P, Pichi A, Laghi A. Bowel cleansing before CT colonography: comparison between two minimal-preparation regimens. Eur Radiol. 2015 Jan;25(1):203-10. doi: 10.1007/s00330-014-3345-0. Epub 2014 Aug 23. PMID 25149295